CLINICAL TRIAL: NCT04243109
Title: Pilot Study (Phase II) of Pomalidomide, Oral Dexamethasone and Very Low-dose Cyclophosphamide in Patients With Refractory Multiple Myeloma Who Have Received Lenalidomide and Bortezomib
Brief Title: Study of Pomalidomide, Oral Dexamethasone and Very Low-dose Cyclophosphamide in Patients With Refractory Multiple Myeloma Who Have Received Lenalidomide and Bortezomib
Acronym: POCODEX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate. Lack of interest of the sponsor.
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCO-PDC-2015-01
Record Dates: First submitted 2019-11-11; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Pomalidomide; Cyclophosphamide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide + Cyclophosphamide + Dexamethasone (Experimental): Treatment Phase: Combination of Pomalidomide, Cyclophosphamide and Dexamethasone, days 1-21 every 4 weeks (28 day cycles), up to a total of 8 cycles:
  * Pomalidomide: Treatment with Pomalidomide 4 mg / day 1-21 days in 28-day cycles is started.
  * Cyclophosphamide: Cyclophosphamide will be administered 15 mg / day, days 1-28 in 28-day cycles.
  * Dexamethasone: Dexamethasone will be administered 40 mg / day, days 1, 8, 15 and 22 in 28-day cycles.
  Maintenance Phase: Combination of Pomalidomide and Dexamethasone. The last doses prescribed in the previous cycle will be maintained.
  Interventions: Drug: Pomalidomide + Cyclophosphamide + Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide + Cyclophosphamide + Dexamethasone — Treatment Phase: Combination of Pomalidomide, Cyclophosphamide and Dexamethasone, days 1-21 every 4 weeks (28 day cycles), up to a total of 8 cycles:
  * Pomalidomide: Treatment with Pomalidomide 4 mg / day 1-21 days in 28-day cycles is started. Dose reductions will be made based on the evaluation of hematological and non-hematological toxicity.
  * Cyclophosphamide: Cyclophosphamide will be administered 15 mg / day, days 1-28 in 28-day cycles.
  * Dexamethasone: Dexamethasone will be administered 40 mg / day, days 1, 8, 15 and 22 in 28-day cycles. In patients older than 75 years the dose will be reduced to 20 mg / day in the same previous schedule.
  Maintenance Phase: Combination of Pomalidomide and Dexamethasone. The last doses prescribed in the previous cycle will be maintained.

SUMMARY:
Clinical trial with a pharmaceutical specialty in a new combination.

Pomalidomide in combination with dexamethasone is indicated in the treatment of adult patients with multiple treatment-resistant or relapsing myeloma who have received at least two previous treatments, including lenalidomide and bortezomib, and who have experienced a disease progression in the last treatment.

The combination of Pomalidomide with Cyclophosphamide at metronomic doses (Very low doses) and Dexamethasone is tested in this clinical situation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age and who meets criteria 2 and / or 3.
* Patient diagnosed with symptomatic Multiple Myeloma according to standard criteria.
* Patients with symptomatic multiple myeloma in relapse / refractory after having received treatment with at least two cycles that include Bortezomib and with at least two cycles that include Lenalidomide, whether combined in the same therapeutic scheme or as part of different chemotherapy schemes.
* Patients with MM with measurable disease, defined as the presence of monoclonal component of at least 0.5 g / dL in serum or at least 0.2 g / d in urine, or in those without measurable disease the presence of altered light chain radius at the time of entry into the study.
* Patients with good general condition defined as ECOG ≤ 2.
* The patient must understand the written informed consent and sign it of his own accord.
* The patient must be able to meet all scheduled visits and other requirements.
* Laboratory Criteria: Patients must present the following counts:Absolute neutrophils: ≥1000 / μL, Platelet Count: ≥50,000 / μL, Hemoglobin:> 8 gr / dL, Total bilirubin: <2 x upper limit of normal, AST and ALT: <3 x Upper limit of normal, Serum potassium: within the limits of normality.
* Women of childbearing age should have a negative pregnancy test.
* The male patient included in the trial must commit to always use a latex condom during any sexual contact with women of childbearing age, even if they have undergone a successful vasectomy.

Exclusion Criteria:

* Any concomitant disease, laboratory alteration or psychiatric disorder that may presuppose the subject's inability to sign the IC.
* PS> 3 according to the ECOG scale.
* Previous history of non-hematologic malignancies, unless the patient has been free of the disease for ≥ 5 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast.
* Patients who are unable or unwilling to undergo antithrombotic therapy.
* Known positive serology for human immunodeficiency virus HIV or active infectious hepatitis, type B, or C.
* Depressed heart function, or clinically significant heart disease
* Severe hypercalcemia
* Major surgical interventions within 15 days prior to inclusion or not having recovered from their side effects.
* Any serious medical condition, including laboratory alterations that cause the patient to take an unacceptable risk if participating in this study or that may interfere with the interpretation of the study data.
* Patients treated with any investigational drug in the previous 28 days.
* Any severe medical condition, abnormality in laboratory tests or any psychiatric illness that prevents the signing of written consent.
* Pregnant or breastfeeding women.
* Known hypersensitivity to drugs or compounds of biological or chemical composition similar to those of the study.
* Plasma Cell Leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Best response | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  Evaluate the best response rate based on the criteria of the International Myeloma Working Group of the following responses at the end of each cycle or during the maintenance period.

SECONDARY OUTCOMES:
Time to Response | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  From the entry into the study or the start of treatment until the first evidence of a confirmed response.
Duration of Response | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  Time from the first evidence of response to the progression or recurrence of the disease.
Time to Progression | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  From the entry into the study or the start of treatment to the progression or recurrence of the disease.
Global Survival | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  from the entry into the study or the start of treatment until the date of death of the patient or the last date on which it was known that the patient was alive.
Progression Free Survival | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  from the entry into the study or the start of treatment to the progression or recurrence of the disease (includes death from myeloma)
Tolerability of the study medication | Every 28 days (each cycle is 28 days) from randomization until progression or withdrawal of the subject, whichever came first, assessed up to 60 months.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0.
Angiogenesis markers of metronomic chemotherapy activity | At baseline and before the beginning of the 2nd, 4th, 6th and 8th treatment cycle (each cycle is 28 days)
  Evaluations of treatment of Circulating Endothelial Cells by multiparameter flow cytometry.
Angiogenesis markers of metronomic chemotherapy activity 2 | At baseline and before the beginning of the 2nd, 4th, 6th and 8th treatment cycle (each cycle is 28 days)
  Evaluations of treatment of Circulating Endothelial Cells by serum levels of VEGF, TSP1.
Immune system evaluation of metronomic chemotherapy activity | At baseline and before the beginning of the 2nd, 4th, 6th and 8th treatment cycle (each cycle is 28 days)
  Evaluation of the Immune system by the determination of regulatory T populations.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel Álvarez Rivas, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available.
  Individual participant data that underlie the results reportes in this article, after deidenttification (text, tables, figures and appendices)
  The other documents that will be available: study protocol, Statistical Analysis Plan, Informed Consent Form.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Open, under previous request.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.